CLINICAL TRIAL: NCT00237679
Title: Quantifying Effects of Treatment of Pediatric Dysphonia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated due to funding loss.
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institute on Deafness and Other Communication Disorders (NIDCD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000-487; R03DC005917 (NIH)
Record Dates: First submitted 2005-10-07; First posted 2005-10-12 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2015-10

CONDITIONS: Voice Disorders; Gastroesophageal Reflux
Keywords: behavior therapy; combination therapy; gastrointestinal disorder chemotherapy; human therapy evaluation; larynx disorder; middle childhood (6-11); lansoprazole; reflux esophagitis; quality of life; clinical research; human subject; laryngoscopy; patient oriented research; questionnaire
MeSH Terms: conditions — Voice Disorders; Gastroesophageal Reflux; Laryngeal Diseases; Esophagitis, Peptic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Neuromuscular Electrical Stimulation (Active Comparator): Subjects will receice Neuromuscular Electrical Stimulation (NMES)-stimulated swallowing combined with exercise therapy.
  Interventions: Behavioral: Neuromuscular Electrical Stimulation
- Unstimulated (Sham Comparator): Subjects will receive sham (unstimulated) swallow therapy combined with exercise therapy.
  Interventions: Behavioral: Unstimulated

INTERVENTIONS:
Behavioral: Neuromuscular Electrical Stimulation — Through low voltage current delivered through the skin, motor nerves are excited, causing muscle contraction.
  Arms: Neuromuscular Electrical Stimulation
Behavioral: Unstimulated — No current is generated.
  Arms: Unstimulated

SUMMARY:
The diagnosis and management of childhood dysphonia is a significant clinical problem; however, there have been few studies aimed at defining standard assessment methods for pediatric dysphonia. Accordingly, pediatric dysphonia is difficult to diagnose and it is difficult to quantify change following treatment. The long-term goal of this research program is to develop valid, responsive, reliable, and age-appropriate methods for assessing vocal pathology in children. In the present small grant, our objective is to define assessment methods that are appropriate for use in determining response to treatment. Our main focus, therefore, is the issue of assessment responsivity. The first specific aim is to develop a set of responsive measures of vocal pathology in school-aged children by inducing short-term change in vocal status via behavioral and medical management of extraesophageal reflux disease (EERD). Because we are treating children suspected of EERD, this study also presents the opportunity for examining the benefits of combined vocal hygiene and medical management in the treatment of pediatric EERD. Accordingly, our second specific aim is to determine predictive criteria for improvement in vocal status in dysphonic children suspected of EERD. Our hypothesis is that a particular set of measurements will emerge as particularly responsive to change in vocal pathology in this population, and will allow for informed prediction of degree of improvement with treatment. The proposed research is significant in filling a gap in knowledge in childhood dysphonia assessment and treatment, which are important clinical issues consistent with the mission and intent of the NIDCD. Because phonatory disorders in children may have lasting negative effects, studies geared toward accurate assessment and treatment are very important.

ELIGIBILITY:
Inclusion Criteria:

* chronic dysphonia with suspected extraesophageal reflux

Exclusion Criteria:

* previous reflux treatment.
* laryngeal disorder treated primarily with surgery

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2004-01; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Determine the effectiveness of medical treatment for hypopharyngeal EERD in dysphonic children. | 3 years
  Determine the effectiveness of medical treatment for hypopharyngeal EERD in dysphonic children.

CONTACTS AND LOCATIONS:
Overall Officials: J. Scott McMurray, MD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin, Madison, Wisconsin, United States